CLINICAL TRIAL: NCT04958759
Title: The Effects of Functional Inspiratory Muscle Training on Respiratory and Peripheral Muscle Functions in Chronic Kidney Disease
Brief Title: Functional Inspiratory Muscle Training in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20086
Record Dates: First submitted 2021-05-12; First posted 2021-07-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Respiratory muscle
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional Inspiratory Muscle Training Group (Experimental): Functional inspiratory muscle training in patients with chronic kidney disease
  Interventions: Other: Functional Inspiratory Muscle Training; Other: Inspiratory Muscle Training
- Inspiratory Muscle Training Group (Experimental): Inspiratory muscle training in patients with chronic kidney disease
  Interventions: Other: Inspiratory Muscle Training
- Control Group (Experimental): Breathing exercises in patients with chronic kidney disease
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training — The inspiratory muscle training program will be consist of 4 weeks of foundation inspiratory muscle training and 6 weeks of functional inspiratory muscle training
  Arms: Functional Inspiratory Muscle Training Group
Other: Inspiratory Muscle Training — The inspiratory muscle training program will be consist of 10 weeks of foundation inspiratory muscle training
  Arms: Functional Inspiratory Muscle Training Group; Inspiratory Muscle Training Group
Other: Breathing exercises — The program will be consist of 10 weeks of breathing exercises
  Arms: Control Group

SUMMARY:
Effects of functional inspiratory muscle training by telerehabilitation on respiratory and peripheral functions, functional capacity, diaphragm thickness and mobility, posture, quality of life, cognitive function, fatigue, physical activity, endothelial function and aortic stiffness in patients with chronic kidney disease will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease not receiving dialysis
* Access to the online program
* Volunteering to participate in the research

Exclusion Criteria:

* Having a musculoskeletal problem
* Having decompensated diabetes
* Having uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 10 minutes
  Respiratory muscle strength will be evaluated using mouth pressure device
Respiratory muscle endurance | 10 minutes
  Respiratory muscle endurance will be evaluated using incremental load test
Pulmonary function | 5 minutes
  Pulmonary functions will be evaluated using spirometry
Peripheral muscle strength | 5 minutes
  Peripheral muscle strength will be evaluated using dynamometer
Endurance of trunk muscles | 10 minutes
  Endurance of trunk muscles will be evaluated using plank, side plank, flexor endurance and pelvic bridge test
Lower extremity muscle endurance | 1 minutes
  Lower extremity muscle endurance will be evaluated using sit-to-stand test
Functional capacity | 10 minutes
  Functional capacity will be evaluated using six-minute walk test
Diaphragm thickness and mobility | 20 minutes
  Diaphragm thickness and mobility will be evaluated using ultrasonography

SECONDARY OUTCOMES:
Balance | 5 minutes
  Balance will be evaluated using timed up and go test
Static balance | 5 minutes
  Balance will be evaluated using one-legged standing test
Posture | 5 minutes
  Posture will be evaluated using Corbin Postural Assessment scale. Lateral and posterior views will be assessed (0 = absent, 1 = mild, 2 = moderate, 3 = severe) and posture score will be determined as excellent (0-2), very good (3-4), good (5-7), fair (8-11) and poor (>12).
Qol | 10 minutes
  Quality of life will be evaluated using Nottingham Health Profile
Cognitive function | 5 minutes
  Cognitive function will be evaluated using Standardised Mini-Mental State Examination
Fatigue | 5 minutes
  Fatigue will be evaluated using Multidimensional Assessment of Fatigue scale
Physical activity | 5 minutes
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short Form
Endothelial function | 10 minutes
  Endothelial function will be evaluated using echocardiography. After a resting baseline Brachial artery diameter will be recorded, the cuff used in blood pressure measurement will be inflated 25-50 mmHg above the systolic blood pressure value and maintaining that pressure for 5 min. The brachial artery diameter will be measured again after the cuff is deflated.
Aortic stiffness | 10 minutes
  Aortic stiffness will be evaluated using transthoracic echocardiography. Aortic diameters can be measured by M-mode tracing of the level of 3-4 cms above the aortic valve during diastole and systole

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, MSc, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Tolga Yildirim, MD, Study Director — Hacettepe University; Deniz İnal-İnce, Professor, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik-Kutukcu, PhD, Study Chair — Hacettepe University; Ahmet Hakan Ates, MD, Study Chair — Hacettepe University; Selin Ardali-Duzgun, MD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)